CLINICAL TRIAL: NCT00058071
Title: A Randomized Phase III Trial of Amifostine vs. No Treatment for Platinum Induced Peripheral Neuropathy
Brief Title: Amifostine in Treating Peripheral Neuropathy in Patients Who Have Received Chemotherapy for Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000285700; GOG-0192
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2007-07

CONDITIONS: Gestational Trophoblastic Tumor; Neurotoxicity; Peripheral Neuropathy; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: peripheral neuropathy; neurotoxicity; hydatidiform mole; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Gestational Trophoblastic Disease; Neurotoxicity Syndromes; Peripheral Nervous System Diseases; Hydatidiform Mole | interventions — Amifostine

INTERVENTIONS:
Drug: amifostine trihydrate

SUMMARY:
RATIONALE: Amifostine may be effective in relieving numbness, tingling, and other symptoms of peripheral neuropathy. It is not yet known whether amifostine is effective in treating peripheral neuropathy in patients who have received chemotherapy for cancer.

PURPOSE: This randomized phase III trial is studying amifostine to see how well it works compared to observation in relieving numbness, tingling, and other symptoms of peripheral neuropathy in patients who have received platinum-based chemotherapy (such as cisplatin or carboplatin) for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine, preliminarily, whether amifostine is superior to no treatment, in terms of improving the symptoms and/or objective findings of platinum-induced peripheral neuropathy, in patients with cancer.
* Determine the toxicity of this drug in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive amifostine IV or subcutaneously over 3 minutes on days 1, 3, and 5. Treatment continues for 12 weeks in the absence of unacceptable toxicity. Patients are observed for 12 weeks.
* Arm II: Patients are observed for 24 weeks. After 24 weeks patients may cross over to treatment as in arm I.

Quality of life is assessed at baseline and then at 6, 12, 18, and 24 weeks after study entry.

Patients are followed at 6 and 12 weeks after study treatment, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 50-100 patients (25-50 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Prior therapy with platinum-based chemotherapy regimen for a malignancy

  * Treatment with other agents, including paclitaxel, allowed
* Grade 2 or greater peripheral neuropathy (numbness, tingling, pain in the distal extremities) attributed to prior platinum-based chemotherapy

  * Must have persisted and be stable for 3-36 months after completion of chemotherapy
  * Duration of neuropathy no more than 3 years
* No other possible causes for the neuropathy (e.g., alcoholism, diabetes, or peripheral vascular disease)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* GOG 0-3

Life expectancy

* At least 6 months

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 2.0 mg/dL

Renal

* Creatinine no greater than 2.0 mg/dL
* Calcium at least lower limit of normal

Cardiovascular

* No hypotension
* No history of cerebrovascular accident

Other

* No other significant comorbid medical conditions that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No concurrent chemotherapy
* No chemotherapy (including paclitaxel, cisplatin, and carboplatin) for at least 4 months after study entry

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 24 hours since prior antihypertensive medications
* No prior amifostine
* Prior treatment on a GOG treatment protocol allowed
* No concurrent monoamine oxidase inhibitors
* No concurrent neurotoxic agents during and for at least 6 months after study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2003-03; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Improvement of neuropathy by WEST assessment at 6, 12, 18, and 24 weeks

SECONDARY OUTCOMES:
Improved quality of life by Functional Assessment of Cancer Therapy-GOG/NTX (FACT-GOG/NTX) at 6, 12, 18, and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Steven C. Plaxe, MD, Study Chair — University of California, San Diego
Locations (57):
- United States (57):
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Moores UCSD Cancer Center, La Jolla, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - St. Vincent's Medical Center, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital at Howard Regional Health System, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Louisville Oncology at Norton Cancer Center, Louisville, Kentucky
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Women's Cancer Center - Lake Mead, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Cancer Care Associates - Midtown Tulsa, Tulsa, Oklahoma
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota